CLINICAL TRIAL: NCT04019431
Title: Very Low-calorie Ketogenic Diet (VLCKD) Influences Taxonomic Composition of the Gut Microbiota and Visceral Adipose Tissue Distribution in Obese Patients With Type 2 Diabetes or Prediabetes Depending on Protein Source
Brief Title: Effect of a Very Low-Calorie Ketogenic Diet on Gut Microbiota and Fat Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1236-5158
Record Dates: First submitted 2019-07-05; First posted 2019-07-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Whey Proteins; Plant Proteins, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein (Experimental): VLCKD (780 kcal/day) low in carbohydrates (<50 g per day) and lipids (only 10 g of olive oil per day) for 45 days. High-biological-value protein preparations will be given four times per day, based on whey protein.
  Interventions: Dietary Supplement: Whey protein, vegetable protein or animal protein
- Vegetable proteins (Active Comparator): VLCKD (780 kcal/day) low in carbohydrates (<50 g per day) and lipids (only 10 g of olive oil per day) for 45 days. High-biological-value protein preparations will be given four times per day, based on vegetal protein derived from soya or green peas or cereals.
  Interventions: Dietary Supplement: Whey protein, vegetable protein or animal protein
- Animal proteins (Active Comparator): VLCKD (780 kcal/day) low in carbohydrates (<50 g per day) and lipids (only 10 g of olive oil per day) for 45 days.Patients will be given four meals per day containing natural animal protein (meat, fish, eggs, dairy products without whey protein).
  Interventions: Dietary Supplement: Whey protein, vegetable protein or animal protein

INTERVENTIONS:
Dietary Supplement: Whey protein, vegetable protein or animal protein — meal replacements or animal protein

SUMMARY:
Short-term interventions that use very low-calorie ketogenic diets and meal replacements may be prescribed for selected overweight or obese patients with type 2 diabetes or prediabetes. Few, inconsistent data are available on protein intake from various sources on body weight, the composition of gut microbiota and metabolic outcomes in these patients. The aim of the present study is to compare efficacy, safety and effect on microbiota composition of short-term isocaloric VLCKDs using whey proteins, vegetable proteins or animal proteins in obese patients with diabetes or prediabetes. 50 obese diabetic/prediabetic patients will be randomly assigned to three isocaloric VLCKD regimens (≤800 kcal/day) containing either whey, plant or animal proteins for 45 days. Outcome measures will be anthropometric parameters, vital signs, metabolic profile, body composition and microbiota assessment.

DETAILED DESCRIPTION:
Short-term interventions that use very low-calorie ketogenic diets and meal replacements may be prescribed for selected overweight or obese patients with type 2 diabetes or prediabetes. Few, inconsistent data are available on protein intake from various sources on body weight, the composition of gut microbiota and metabolic outcomes in these patients. The aim of the present study is to compare efficacy, safety and effect on microbiota composition of short-term isocaloric VLCKDs using whey proteins, vegetable proteins or animal proteins in obese patients with diabetes or prediabetes. 50 obese diabetic/prediabetic patients will be randomly assigned to three isocaloric VLCKD regimens (≤800 kcal/day) containing either whey, plant or animal proteins. Outcome measures will be anthropometric parameters, vital signs, metabolic profile, body composition and microbiota assessment. The patients will be assessed at baseline (T0) and every two weeks (T15, T30) up to day 45 (T45) when they will be finally evaluated. Patients will be given support and counselling to enhance their compliance. The patients will also be instructed to have moderate-intensity physical activity (e.g., 30 minutes walking every day) during the study.

Anthropometric parameters Body weight, blood pressure (systolic and diastolic), heart rate, waist and hip circumference will be measured at baseline (T0), every two weeks up to the end of the trial (T45).

Blood and urine chemistry Complete Blood Count (CBC), electrolytes (chloride, calcium, potassium, sodium, magnesium), fasting glucose, insulin, lipids (total and fractionated cholesterol and triglycerides) and proteins, C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), plasma creatinine, blood urea nitrogen (BUN), alanine transferase (AST), aspartate transaminase (ALT), uric acid and estimated Glomerular Filtration Rate (using the Modification of Diet in Renal Disease study equation MDRD-eGFR) will be determined at baseline and after 45 days.

The overnight fasting plasma levels of Insulin Like Growth Factor-1 (IGF-1) will be measured using commercially available ELISA kits. Urine tests will be performed at baseline and every other week until the end of the study.

Dual-Energy-X-ray Absorptiometry measurement (DEXA) Body composition, total and regional body fat mass (FM) and fat-free mass (FFM), will be measured using DEXA (Hologic 4500 RDR) at baseline and at the end of the trial.

Visceral adipose tissue (VAT) will be calculated using a fully automated software. DEXA-VAT will be measured in a 5 cm wide area placed in the abdominal region just above the iliac crest, at a level that approximately coincides with the 5th lumbar vertebrae on the whole body DEXA scan. The VAT will be estimated by subtracting subcutaneous fat from the total abdominal fat by means of an algorithm.

Muscular strength Muscle strength will be measured through a digital dynamometer handgrip at T0 and T45. Before starting, patients will be asked to squeeze as hard as possible the dynamometer for at least 3 seconds. Three measurements will be repeated with both the dominant and non-dominant arms. The highest value measured will be recorded as the maximum grip force.

Taxonomic composition of the gut microbiome Fecal sampling will be done using sterile swab and tubes DNA purity will be evaluated based on A260/A280 ratio using a spectrophotometer. DNA integrity and size will be assessed by 1.5% agarose gel electrophoresis. The V3-V4 region of the 16S ribosomal RNA gene will be amplified. Polymerase Chain Reaction (PCR) amplicons will be purified and amplified following the Nextera XT Index protocol. The processed reads will be clustered and the operational taxonomic units will be assigned to taxa.

Data obtained will be expressed as mean values ±Standard Deviation (SD) and finally processed to ascertain whether statistical differences among them can be demonstrated, using appropriate methods. In particular, the analysis of variance (ANOVA) at different times will be used for efficacy and safety data, such as weight reduction, changes in anthropometric measures, FM and FFM and variation of the metabolic parameters. P values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI 30-40)
* newly-diagnosed and untreated type 2 diabetes (fasting plasma glucose ≥ 126 mg/dL or HbA1c ≥ 6.5 mmol/L) or impaired fasting glycemia (fasting plasma glucose from 110mg/dl to 125mg/dl).
* stable body weight in the previous 3 months

Exclusion Criteria:

known hypersensitivity to one or more components used in the protocol products; history of renal, cardiac, cerebrovascular or gastrointestinal diseases; psychiatric disturbances; hydroelectrolytic alterations, diagnosis of type 1 diabetes lack of informed consent; history of or planned weight loss surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index change from baseline | 45 days
  Body Mass Index will be calculated at baseline and after 45 days

SECONDARY OUTCOMES:
Fat mass percentage (%) change from baseline | 45 days
  Fat mass percentage will be assessed by DXA at baseline and after 45 days
Visceral adipose tissue (gr) change from baseline | 45 days
  Visceral adipose tissue will be assessed by DXA at baseline and after 45 days
Microbiome taxonomic composition change from baseline | 45 days
  Change in abundance of gut microbiome will be measured with stool sample collections at baseline and after 45 days
Fasting glucose level (mg/dL) change from baseline | 45 days
  blood glucose will be measured at baseline and after 45 days
Fasting Insulin level (mcU/mL) change from baseline | 45 days
  insulin will be measured at baseline and after 45 days
Fasting Cholesterol level (mg/dL) change from baseline | 45 days
  Fasting Cholesterol will be measured at baseline and after 45 days
Muscle strength (kg) change from baseline | 45 days
  Muscle strength will be assessed with a handgrip test at baseline and after 45 days
Quality of life (subjective unit) change from baseline | 45 days
  Quality of life will be assessed through questionnaire
Safety (subjective unit) change from baseline | 45 days
  safety will be assessed through questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Gnessi, MD PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basciani S, Camajani E, Contini S, Persichetti A, Risi R, Bertoldi L, Strigari L, Prossomariti G, Watanabe M, Mariani S, Lubrano C, Genco A, Spera G, Gnessi L. Very-Low-Calorie Ketogenic Diets With Whey, Vegetable, or Animal Protein in Patients With Obesity: A Randomized Pilot Study. J Clin Endocrinol Metab. 2020 Sep 1;105(9):dgaa336. doi: 10.1210/clinem/dgaa336. PMID 32484877